CLINICAL TRIAL: NCT01964482
Title: In-hospital and Post-discharge Training of Older Medical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Mette Merete Pedersen, PhD student, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2-2012-115
Record Dates: First submitted 2013-10-14; First posted 2013-10-17 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Hospitalized Older Medical Patients
Keywords: Hospitalization; Older; Medical patient; Strength training
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Strength training (Experimental): Supervised strength training daily during hospitalization and 3 times per week for 4 weeks after discharge in the participant's home
  Interventions: Other: Strength training
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Other: Strength training — Strength training followed by intake of a protein drink
  Arms: Strength training

SUMMARY:
The project aims to investigate the clinical value of simple strength training during hospitalization and after discharge as part of an enhanced recovery programme for acutely admitted older medical patients, in order to prevent mobility decline following acute hospitalization.

Note 11/23/16: As noted in the protocol (doi: 10.1186/s13063-016-1309-1) we have obtained funding and ethical approval (H-2-2012-115/09-12-2016) to extend the study to achieve sufficient power to look more deeply into our secondary outcomes. This will constitute a secondary part of the trial (started Nov. 2016). The primary trial report will include data for the pre-specified sample size for which the last patient was assessed Oct. 2016. Hence, the primary completion date for part 1 was April 2016 and the study completion date for part 1 was Oct 2016. The trial status is still "recruiting" although this applies to part 2 of the study.

ELIGIBILITY:
Inclusion Criteria:

* >=65 years of age
* admitted from own home

Exclusion Criteria:

* Terminal illness
* In treatment for diagnosed cancer
* Assigned to physical rehabilitation in community
* Chronic Obstructive Pulmonary Disease (COPD) patients participating in organized rehabilitation
* Living outside of the municipalities of Copenhagen and Broendby
* Not able to talk and understand danish
* Not able to cooperate on tests/exercises
* Hospitalized < 24 hours
* A Cumulated Ambulation Score (CAS) of 0 in the sit-to-stand item

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 158 (Actual)
Dates: Start 2013-10; Primary Completion 2016-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Mobility using the de Morton Mobility Index (DEMMI) | Admittance (baseline), discharge, 4 weeks after discharge (primary analysis), and 26 weeks after discharge
  The DEMMI is an advanced instrument for accurately measuring the mobility of older people across clinical settings (www.demmi.org.au). The primary analysis for the primary outcome is the change in the DEMMI score from baseline to the assessment 4 weeks after discharge (end of intervention). The primary analysis will follow the intention-to-treat principle (last observation carried forward) and be unadjusted in order to determine a systematic group-difference in the change from baseline to 4 weeks post discharge (end of training) for the primary outcome.

SECONDARY OUTCOMES:
Isometric knee-extension strength in dominant leg | At admittance (baseline), at discharge, 4 weeks after discharge and 26 weeks after discharge
  Isometric knee-extension strength will be measured using an externally fixated handheld dynamometer (Power Track II Commander; JTech Medical, Utah). A stap will be attached to the bed/chair and the patient's ankle (perpendicular to the lower leg), ensuring 90 degrees of knee flexion and an isometric contraction. The transducer will be placed under the strap at ankle level, just proximal to the malleolus, and the participant will be asked to extend the leg as forcefully as possible. Knee-extension strength will be expressed as the maximal voluntary torque per kilo body mass ([NIm]/kg), using the distance between the lateral femoral epicondyle and the center of the transducer and the body mass of each patient.
Hand-grip strength of dominant hand | Admittance (baseline), discharge, 4 weeks post discharge and 26 weeks post discharge
  Isometric handgrip strength will be measured in the dominant hand using a handheld dynamometer (Digi-II; Saehan). The patient will be placed in a sitting position in an armchair, with the lower arm placed on the arm rest and an elbow flexion of 90 degrees. The patients will be asked to squeeze the handle as forcefully as possible for 5 secs. Handgrip strength will be expressed in kilograms.
30-sec sit to stand test | Admittance (baseline), discharge, 4 weeks post discharge, 26 weeks post discharge
  The patients will be asked to stand up and sit down as many times as possible in 30 secs with their arms across their chest.
Habitual gait speed | Admittance (baseline), discharge, 4 weeks post discharge, 26 weeks post discharge
  Patients will be asked to walk a 4-meter straight walk at their usual pace starting from a standing position.
24-hour mobility | Admittance to discharge, discharge to 1 week post discharge, 4 weeks post discharge to 5 weeks post discharge, 26 weeks post discharge to 27 weeks post discharge (4 x 1 week)
  The patients will be asked to wear an ActivPAL3 activity monitor (PAL Technologies Ltd, Scotland) on the thigh during hospitalization, the first week after discharge, the first weeks after the 4-week assessment and the first week after the 26-week assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Mette M Pedersen, PhD Student, Principal Investigator — Hvidovre Hospital, University of Copenhagen; Thomas Q Bandholm, PhD, Study Director — Hvidovre Hospital, University of Copenhagen; Janne Petersen, PhD, Study Director — Hvidovre Hospital, University of Copenhagen
Locations (1):
- Copenhagen University Hospital, Hvidovre, Hvidovre, Denmark

REFERENCES:
- [Derived] Bornaes O, Andersen AL, Houlind MB, Kallemose T, Tavenier J, Aharaz A, Nielsen RL, Jorgensen LM, Beck AM, Andersen O, Petersen J, Pedersen MM. Mild Cognitive Impairment Is Associated with Poorer Nutritional Status on Hospital Admission and after Discharge in Acutely Hospitalized Older Patients. Geriatrics (Basel). 2022 Sep 10;7(5):95. doi: 10.3390/geriatrics7050095. PMID 36136804
- [Derived] Pedersen MM, Petersen J, Beyer N, Larsen HG, Jensen PS, Andersen O, Bandholm T; STAND-Cph collaborative group. A randomized controlled trial of the effect of supervised progressive cross-continuum strength training and protein supplementation in older medical patients: the STAND-Cph trial. Trials. 2019 Nov 28;20(1):655. doi: 10.1186/s13063-019-3720-x. PMID 31779693
- [Derived] Pedersen MM, Petersen J, Beyer N, Damkjaer L, Bandholm T. Supervised progressive cross-continuum strength training compared with usual care in older medical patients: study protocol for a randomized controlled trial (the STAND-Cph trial). Trials. 2016 Apr 1;17:176. doi: 10.1186/s13063-016-1309-1. PMID 27039381